CLINICAL TRIAL: NCT07002580
Title: Evaluation of the Effectiveness of iPACK (Local Anesthetic Infiltration of the Interspace Between the Popliteal Artery and the Posterior Knee Capsule) and Adductor Canal Blocks on Quality of Recovery in Patients Undergoing Arthroscopic Knee Surgery
Brief Title: Evaluation of the Effectiveness of iPACK and Adductor Canal Blocks on Patients Undergoing Arthroscopic Knee Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Oguzhan Okumus, Resident M.D., Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-43012747-050.04-463720-202
Record Dates: First submitted 2025-05-15; First posted 2025-06-03 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-05

CONDITIONS: Patients Undergoing Arthroscopic Knee Surgery
Keywords: Arthroscopic Knee Surgery; Perifheric Nerve Block; Analgesia; iPACK; Adductor Canal Block; QoR-15
MeSH Terms: conditions — Agnosia | interventions — Anesthesia, Spinal; Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients will be randomized with closed letter method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Group 1 will involve the patients which will be applied iPACK and adductor canal blocks in addition to spinal anesthesia.
  Interventions: Procedure: IPACK and adductor canal block with Bupivacaine 0.25%; Procedure: Spinal Anesthesia with Bupivacaine
- Group 2 (Experimental): Group 2 will involve the patients which will be applied only spinal anesthesia without additional peripheric nerve blocks.
  Interventions: Procedure: Spinal Anesthesia with Bupivacaine

INTERVENTIONS:
Procedure: IPACK and adductor canal block with Bupivacaine 0.25% — iPACK block is infiltration between the Popliteal Artery and the Capsule of the Knee. iPACK and adductor canal blocks are performed with ultrasound guidence under sterile conditions.
  Arms: Group 1
Procedure: Spinal Anesthesia with Bupivacaine — Spinal Anesthesia is a basic anesthesia method used for years to grant anesthesia for surgeries for lower extremities and lower torso surgeries.

SUMMARY:
Arthroscopic knee surgery is one of the most commonly performed procedures in orthopedic surgery. More than 50% of patients experience moderate to severe pain after the operation. Inadequate postoperative pain control and poor recovery quality can negatively impact physiotherapy protocols, prolong hospital stays, and consequently lead to cognitive dysfunction, systemic infections, and increased healthcare costs.

Therefore, reducing postoperative pain and improving recovery quality are of great importance. In our clinic, a variety of analgesic techniques are routinely employed as part of a multimodal analgesia approach for patients undergoing arthroscopic knee surgery. One of these techniques is the simultaneous application of the IPACK block and the adductor canal block.

In this study, we aim to evaluate the effectiveness of these blocks on postoperative recovery quality in patients undergoing arthroscopic knee surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 50 years,
* Scheduled for arthroscopic knee surgery under spinal anesthesia due to knee pathology
* Patients classified as ASA physical status I-II-III according to the American Society of Anesthesiologists risk classification

Exclusion Criteria:

* Coagulopathy
* ASA IV-V patients
* Uncooperable patients
* Patients who refuses to participate in study
* Patients who takes chronic pain treatments

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-01-01 (Actual); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Quality of Recovery | 24 hours.
  Quality of Recovery of the patients will be assessed with QoR-15 questionnaire. Its scoring will range between 0 and 150 points.

SECONDARY OUTCOMES:
Analgesic Consumption | 24 hours.
  The total analgesic consumption of patients according to the patient controlled analgesia device which measures the opioid consumption for 24 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Sakarya University Training and Research Hospital, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided